CLINICAL TRIAL: NCT00511966
Title: Influence of Hygiene-dietetic Habits and Treatment Adherence on the Effectiveness of the Gastroesophageal Reflux Illness Treatment With Rabeprazol
Status: Terminated | Type: Observational
Why Stopped: Due to the achievement of minimum required sample size and new changes in local regulations.
Sponsor: Janssen-Cilag, S.A. (Industry)
Responsible Party: Country Medical Director, Janssen-Cilag S.A., Spain
Other Study IDs: CR009241
Record Dates: First submitted 2007-08-02; First posted 2007-08-06 (Estimated); Last update posted 2011-05-19 (Estimated); Status verified 2010-04

CONDITIONS: Gastroesophageal Reflux
Keywords: Gastroesophageal Reflux; Rabeprazole
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Rabeprazole

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 001
  Interventions: Drug: Rabeprazole
- 002
  Interventions: Other: Non-Pharmacologic Treatment

INTERVENTIONS:
Other: Non-Pharmacologic Treatment — Non-Pharmacologic Treatment
  Groups: 002
Drug: Rabeprazole — As prescribed
  Groups: 001

SUMMARY:
The objective of this Observational study is to evaluate hygiene-dietetic habits as co-adjuvant treatment of the pharmacologic therapy use to treat Gastroesophageal Reflux.

DETAILED DESCRIPTION:
Gastroesophageal Reflux illness is a multifactor pathology with a common mechanism: a prolonged exposure of the esophageal mucosa to the gastric solutions. Modification of the life style and the hygiene-dietetic habits are frequently recommended as an initial therapeutic instrument in Gastroesophageal Reflux pathology. But there is not agreement about the effectiveness of these habits in the improvement of the illness. Different clinical practice guidances have shown contradictions in the effectiveness of changing hygiene-dietetics habits of the life style. The high effectiveness of the new pharmacologic treatment in Gastroesophageal Reflux pathology make it necessary to review the role of hygiene-dietetic habits in this illness. Proton pump inhibitors (PPI) act in the final step of the gastric secretion. PPI's block ATP-ase H+/K+ in gastric parietals cells. This mechanism generates a higher acid inhibition, longer than the inhibition produced by H2-receptor antagonists. It has been described that inhibition of acid secretion has produced a recovery of the gastroesophageal pathology in a high percentage of the patients resistant to conventional drugs. This is an observational, multicenter, open and prospective study. The primary objective is to evaluate hygiene-dietetic habits as co-adjuvant of Rabeprazol treatment in Gastroesophageal Reflux . It is expected to include 570 patients with Gastroesophageal pathology erosive or non-erosive and acute or chronic treated with Rabeprazol per clinical practice, 20mg per day, orally, for 8 weeks. All data collected will be prospective and will include the following: demographic data, progress of the pathology, change of hygiene-dietetic habits, treatment adherence, concomitant treatments and adverse events. Observational Study - No investigational drug administered

ELIGIBILITY:
Inclusion Criteria:

* Patients with Gastroesophageal pathology erosive or non-erosive and acute or chronic treated with Rabeprazol per clinical practice

Exclusion Criteria:

* Patients pregnant or lactating
* Other gastrointestinal pathologies
* Intestinal or gastric survey
* Other severe concomitant pathologies
* Drug abuse or use of NSAIs (Non-Steroidal Anti-Inflammatories) more than 3 days/week

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Gastroesophageal Reflux and symptomatic.
Sampling Method: Non-Probability Sample
Enrollment: 1049 (Actual)
Dates: Study Completion 2002-11 (Actual)

PRIMARY OUTCOMES:
Gastroesophageal Reflux symptoms | 8 weeks

SECONDARY OUTCOMES:
No secondary outcome measures

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag S.A. (formerly Janssen Sp) Clinical Trial, Study Director — Janssen-Cilag, S.A.

REFERENCES:
- See also: Influence of hygiene-dietetic habits and treatment adherence on the effectiveness of the gastroesophageal reflux illness treatment with Rabeprazol. — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=283&filename=CR009241_CSR.pdf